CLINICAL TRIAL: NCT00957255
Title: Rotator Cuff Repair (RCR) With and Without OrthoADAPT Augmentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O-0803
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCR without augmentation (Active Comparator): Rotator cuff repair without OrthoADAPT augmentation
  Interventions: Procedure: Standard of care
- RCR with augmentation (Experimental): Rotator cuff repair with OrthoADAPT augmentation
  Interventions: Device: OrthoADAPT

INTERVENTIONS:
Device: OrthoADAPT — soft tissue augmentation device
  Arms: RCR with augmentation
Procedure: Standard of care — Standard of care rotator cuff repair
  Arms: RCR without augmentation

SUMMARY:
Prospective, randomized, multi-center, controlled study for patients undergoing open rotator cuff repair. Patients are stratified based on tear size to one of three groups. Each group is then randomized 1:1 to either repair with OrthoADAPT or repair without OrthoADAPT.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* MRI confirmed full thickness or high grade partial thickness rotator cuff tear equal or more than 1 cm and involving the supraspinatus and/or infraspinatus tendons
* Tear is repairable by surgery using protocol prescribed fixation procedure
* Patient is able to sign and IRB approved study informed consent
* Patient is willing and able to return for follow-up appointments and study related procedures
* Patient is willing to comply with prescribed physical therapy regimen

Exclusion Criteria:

* Emergency, poly trauma patients
* Prior same shoulder surgery including rotator cuff repair except prior subacromial decompression or distal clavicle resection
* Shoulder pathology requiring concomitant procedures during the rotator cuff repair including Labral repair, anterior or posterior stabilization, and/or capsular plication or shift
* Cervical spine disease
* History of adhesive capsulitis in either shoulder
* Patient whose injury does or may involve litigation
* Diabetics
* Rotator cuff tear cannot be repaired by primary surgical means including superiorly migrated humeral head, retracted rotator cuff that cannot be mobilized to humeral head, end stage tears, rotator cuff tissue cannot retain sutures, any comorbidities that would directly or indirectly affect the reparability of the cuff
* Patients with grade 3 or 4 glenohumeral arthritis
* Patients with systemic collage disease
* Patients with a known hypersensitivity to equine derived materials
* Active or latent infection
* Chronic use of immunosuppressive agents
* Any oral or IM NSAID usage within 5 days before surgery
* Cancer patients
* Decisional impaired patients
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Passive and active range of motion | Pre-op, 6 weeks, 3, 4, 6, 12, and 24 months
American Shoulder and Elbow Surgeons assessment score | Pre-op, 6 weeks, 3, 4, 6, 12, and 24 months
Constant shoulder score | Pre-op, 6 weeks, 3, 4, 6, 12, and 24 months
Pain | Pre-op, 2, 3, 4, and 6 weeks, 3, 4, 6, 12 and 24 months

SECONDARY OUTCOMES:
MRI | 12 months
Rotator cuff re-rupture and adhesions | 6 weeks, 3, 4, 6, 12 and 24 months
Incidence of device or procedure related adverse events | 6 weeks, 3, 4, 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles DePaolo, MD, Principal Investigator — Mission Health Research Institute; Pierce Scranton, MD, Principal Investigator — Seattle Medical Research Foundation; William Bryan, MD, Principal Investigator — Methodist Center for Orthopedic Surgery
Locations (1):
- Seattle Medical Research Foundation, Seattle, Washington, United States